CLINICAL TRIAL: NCT05912920
Title: Laparoscopic Natural Gastric Banding for Management of Morbid Obesity
Brief Title: Laparoscopic Natural Gastric Banding for Morbid Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, prof., Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fac.med 23.25
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gastric band (Experimental): to do gastric banding use either round ligament or omental flap
  Interventions: Procedure: gastric band
- sleeve gastrectomy (Active Comparator): to do sleeve gastrectomy as standard
  Interventions: Procedure: gastric band

INTERVENTIONS:
Procedure: gastric band — gastric band

SUMMARY:
to do gastric banding using round ligament or omental flap instead of synesthetic band

DETAILED DESCRIPTION:
the round ligament or omental flap is used for gastric band instead of synesthetic band which had many complications that led to its abandon

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity
* patients fit for laparoscopic surgery
* give approval to share in the study
* previous restrictive bariatric procedure

Exclusion Criteria:

* patients unfit for surgery
* patients aged less than 18 and older than 60
* patient with previous upper abdominal surgery either for obesity or other diseases

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
%EWL | 12 months
  percentage of excess weight loss at one year

SECONDARY OUTCOMES:
complications rate | 12 months
  the incidence of complications

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of medicine, Minya
  - Minia university hospital, Minya